CLINICAL TRIAL: NCT05389501
Title: Evidence Based Intervention to Improve Social Policy for Maternal and Child Health Using a Pre-Post Test Design
Brief Title: Intervention to Improve Social Policy for Maternal and Child Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Forman Christian College, Pakistan (Other)
Collaborators: UNICEF (Other)
Responsible Party: Principal Investigator, Sara Rizvi Jafree, Associate Professor & Chair, Department of Sociology, Forman Christian College, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 786.NRPU.Social.Policy
Record Dates: First submitted 2022-05-09; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Maternal Health; Maternal Health Literacy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The Experiment Group will receive the following services from the community social worker:
  1. Developing Database on Digital App 2. Community Needs Assessment 3 Pre-Post Test Survey 4. Existing services by government of Pakistan (BHU/ LHW)
  Additionally, the Experiment Group will receive the following services from the health social worker:
  1. Psychosocial needs assessment and mental health awareness
  2. Measurement of Basic Health Clinical Indicators
  33. Health Awareness & Literacy for following areas:
  1. Reproductive and Child Health
  2. Hygiene and Sanitation & Nutrition and Immunity Building
  3. Health-Risk Behavior Modification
  Interventions: Behavioral: Social policy intervention to support women of reproductive years
- Control Group (Active Comparator): The Control Group will receive the following services from the community social worker:
  1. Developing Database on Digital App
  2. Community Needs Assessment 3 Pre-Post Test Survey
  4. Existing services by government of Pakistan (BHU/ LHW)
  Interventions: Behavioral: Social policy intervention to support women of reproductive years

INTERVENTIONS:
Behavioral: Social policy intervention to support women of reproductive years — The project team will attempt to address this challenge by delivering the following interventions through social workers in underdeveloped primary healthcare settings to promote maternal and child health:
  1. Developing a database on a digital app of participants in the study and use the data for development of an Index for Maternal Health and Wellbeing
  2. Conducting a Community Assessment Needs
  3. Conduct a psychosocial needs assessment
  4. Develop interprofessional health workforce collaboration
  5. Measure basic clinical health indicators
  6. Provide health awareness and literacy training to participants

SUMMARY:
Some of the challenges Pakistan faces in priority areas of national relevance include absence of social policy to improve innovative governance and reform of the primary healthcare system, especially for maternal and child health. One integral tool for development of social policy in a country is the integration of the social work profession at primary level. Developed countries have progressed by strengthening the primary workforce with social workers, who have contributed by developing a social policy protection floor for mother and child in primary level communities through: (i) assessment of community needs (e.g. for housing, health, education, and employment), (ii) robust data collection, (iii) political advocacy, and (iv) supporting literacy and counseling . In this way, there is potential to fill a gap by adding Social Workers to the primary health force team in Pakistan to investigate the following research questions:

1. Can a robust, objective, third-party Community Needs Assessment Report (by Social Workers) help to mobilize governments and policy-makers for improve planning and protective policies for disadvantaged communities?
2. Can a more comprehensive health electronic database be developed with both health and social variables to better plan policy development and develop a much-needed regional Index for Maternal Health and Wellbeing?
3. Can maternal and health outcomes be impacted positively by the following intervention this project plans to deliver: (i) Reproductive and Child Health; (ii) Hygiene and Sanitation & Nutrition and Immunity Building; (iii) Health-Risk Behavior Modification; and (iv) Psychosocial Needs Assessment and Mental Health Awareness?
4. Can primary healthcare services become more efficient and effective (in teamwork and improved care plans for client) through interprofessional health workforce collaboration and supplementation of social workers to the team? The proposed project, lasting 24 months, will aid socio-economic development of the country by improving primary healthcare services, improving maternal and child health outcomes, improving preventive behavior overall in families, and strengthening the health workforce team. Improving preventive health also reduces national health costs in the long-run at an estimated USD 45 billion. Building an electronic database with both health and social indicators is integral for the planning of a more effective social and health policy in the future. Integrating social workers at primary level will create thousands of jobs per year for Pakistan and help develop the educations sector as well and provide opportunities for more health workforce development, like public health officers.

The activities that will be undertaken to achieve the project goals include:

1. Development of a digital app and finalization of an Index for Maternal Health and Wellbeing
2. Preparation of a Community Assessment Needs Report for mobilization of social protection floor
3. A Pre-Post Test Survey to measure changes caused by intervention for: (i) Basic Clinical Health Indicators, (ii) Reproductive and Child Health, (iii) Hygiene and Sanitation & Nutrition and Immunity Building, (iv) Health-Risk Behavior Modification; and (v) Psychosocial Assessment and Therapy needs.
4. Dissemination of findings to government bodies, policy-makers, scholars, and researchers to mobilize social policy support and improved governance at primary level through the project pilot model.

An interdisciplinary team of social policy analyst, economist, physician, comprise the main investigators who have developed the proposal and will oversee the study.

They will be supported by a clinical psychologist, biostatistician, and a social statistician for assistance in technical psychosocial assessment and advance data analysis for Pre-Post Test design. Officers from Forman Christian College University will support the project in areas of senior consultancy, IT support and digital app development, and budgeting and audit. Senior consultancy and support for recruitment and training for social workers as data collectors and intervention facilitators will be provided by the University of the Punjab.

The sectoral collaborators and technical consultations, including gaining necessary permissions for data collection in primary settings, will be provided by The Primary & Secondary Healthcare Department, Punjab, Office of the Director General Health Services, Policy & strategic Planning unit (PSPU), development partners (UNICEF, WHO, BMGF), Academia (KEMU) and planning & development department Punjab.

DETAILED DESCRIPTION:
The priority area of national relevance that the project falls under mainly is "Innovative Governance and Reforms", as the target is to improve healthcare governance at primary level and the attempt is to integrate social workers in primary communities, as an integral part of social policy development. Social workers will provide social protection services related to: (i) robust electronic data collection for index development and policy mapping, (ii) assessment of community needs for advocacy for policy development and holding the government to account, and (iii) pre-post test analysis for mediation in literacy, awareness and counseling for local capacity of vulnerable populations (mother and child in underdeveloped communities who are dependent on primary level services for health and social protection). In this way, the project will contribute to innovative solutions for primary health governance strengthening, improvement in preventive health and saving of national health costs in the future, and mobilization for policy reforms for community development. This study will be applied research using direct interventions and thus will contribute to use of open-access data and empirical evidence-based policy design.

In addition the project addresses three other national priority areas as work for social and health policy development is overlapping and cross-cutting, thus benefiting multiple sectors and sub-structures of national relevance. Firstly, the project will include development of an electronic health database through smartphone and digital app, and this will contribute to the priority area of national relevance under "Information Technology and Telecom". The proposed project will contribute to building a robust electronic database using technology, smartphone and 4G Wifi, which will improve Big Data, Index development for assessment and policy design, and scalable models for health and social protection.

Secondly, the project will also include building and integration of social work skills and profession by integrating them in the existing interdisciplinary primary healthcare team and thus contribute to priority area of national relevance under "Development Economics". To be noted is that the existing primary healthcare team (doctors, nurse, and LHW) are overburdened and inefficient. The proposed project will build a case for not just service efficiency in primary health, but add to labor market innovations and demand-side employment for Pakistan.

Lastly, the project through the community assessment of needs will contribute to recommendations for improvement in housing and sanitation, water and food security, waste disposal and sewerage system, transport services, schooling and education services, safety and security, and availability of loan, entrepreneurial and poverty schemes. Recommendations in the report will include suggestions for social protection schemes for improved wellbeing in communities and better planning of underdeveloped or badly managed cities, towns, and villages.

This proposed research is not just important for addressing priority area of national relevance, but also to meet the following five Sustainable Development Goals outlined for developing economies like Pakistan:

(I) SDG 3- Establish Good Health and Well-Being: The project proposes to strengthen primary level services and promote preventive health by delivering interventions for (i) Basic Clinical Health Indicators, (ii) Reproductive and Child Health, (iii)Hygiene and Sanitation & Nutrition and Immunity Building, (iv) Health-Risk Behavior Modification, and (v) Psychosocial Assessment and Therapy needs. It must also be noted that interventions for mothers has direct benefits on self, child and family health and practices. This is timely especially in consideration to the multiple health crises Pakistan faces in communicable and non-communicable diseases and rising health costs.

(II) SDG 5- Enforce Gender Equality: The project proposes to provide efficient and equitable services to target improvement in maternal and child health. The project will directly intervene for improvement in basic clinical health indicators and health awareness and literacy (for Reproductive and Child Health, Hygiene and Sanitation & Nutrition and Immunity Building , and Health-Risk Behavior Modification). It must be noted that newborn and child health is the responsibility of mother, and thus literacy and awareness in women directly children, especially girl children in areas of nutrition and education. It is also known to prevent regressive cultural practices like female feticide and child marriage.

This is timely especially in consideration that Pakistan is facing critical shortfalls in Millennium Development Goal targets for reducing maternal and child mortality.

(III) SDG 10- Reduce Inequality: One component of SDG 10 is reducing inequality between the genders. The study will focus on developing literacy and awareness for women of reproductive years as vulnerable populations. Women in underdeveloped areas that are dependent on primary healthcare services are from the population strata that face inequality issues related to illiteracy or semi-literacy, poverty and unemployment or informal sector employment. Targeting gender equality in health and social service protection for vulnerable populations is timely especially in consideration that the COVID-19 pandemic has directed policy and budget to infection control and health costs as opposed to gender equality.

(IV) SDG 11- Mobilize Sustainable Cities and Communities: The project proposes to provide develop a community needs assessment reports. The benefit of this report will be that it is prepared by the social workers and PIs of the study and as third parties they will provide an objective assessment for policy development and political advocacy. This is timely especially in consideration to the multiple challenges and policy pressures facing the government of Pakistan. Independent research universities must support the government in recommending policy implementation based on empirical evidence and pilot studies.

(V) SDG 17- Build Partnerships for the Goals: The project proposes to build interprofessional health workforce partnership by supplementing existing primary healthcare providers (doctor, nurse an LHW) with social workers (community social worker + health social worker). This will benefit interprofessional collaboration and teamwork for better patient management and development of care plans for patient safety and preventive health. It will also benefit collective policy advocacy to the center by a united primary health workforce. This is timely especially in consideration of the critical challenges facing the existing health workforce at primary level which is overworked, understaffed, inefficient, and unable to collaborate for optimal services and care plans or policy advocacy.

The proposed project is critical because there is very little funding and attention for developing social policy in partnership with health policy. In addition, there is neglect in consideration that research and budget must target preventive health. Currently the Sehat Sahulat Programme is covering mainly hospitalization and has not yet considered service improvement and strengthening of the primary health sector. The project will also aid socio-economic development of the country by improving primary healthcare services, improving maternal and child health outcomes, and improving preventive behavior overall in families, and strengthening the health workforce team. Improving preventive health also reduces national health costs in the long-run at an estimated USD 45 billion. Building of an electronic database and an index for maternal health and wellbeing which includes social indicators can with the planning of more effective social and health policy in the future. Integrating social workers at primary level will create thousands of jobs per year for Pakistan and help develop the educations sector as well and provide opportunities for more health workforce development, like public health officers.

ELIGIBILITY:
Inclusion Criteria:

* Poor women of reproductive years
* Existing clients of doorstep visiting lady health workers (LHWs)

Exclusion Criteria:

- Women not of reproductive years

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 500 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in health literacy of women of reproductive years over 24 months | 2 years
  We will use the standardized international survey: "Knowledge and Reported Practices of Women on Maternal and Child Health" (Kanu, Tang, & Liu, 2014). The following domain areas will be measured including: (i) Pregnancy and antenatal care; (ii) Health knowledge; (iii) Accessing health care; (iv) Vaccinations coverage; (v) Child's father/husband's involvement in maternal and child care; and (vi) Household factors (e.g. hygiene, water and food preparation, waste disposable, and toilet quality, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Kauser R Abdullah Malik, PhD, Study Chair — Forman Christian College, Pakistan
Locations (2):
- Pakistan (2):
  - Forman Christian College University, Lahore, Punjab Province
  - Forman Christian College, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No